CLINICAL TRIAL: NCT03802006
Title: Ultrasound Assessment of Gastric Contents in Fasted Surgical Patients With Previous Subtotal Gastrectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: L-2018-346
Record Dates: First submitted 2019-01-03; First posted 2019-01-14 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2018-10

CONDITIONS: Gastroparesis
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- fasted patient with previous gastrectomy: The fasted patient with previous subtotal gastrectomy except exclusion criteria are included
  Interventions: Diagnostic Test: Ultrasound assessment of gastric content

INTERVENTIONS:
Diagnostic Test: Ultrasound assessment of gastric content — Ultrasound assessment of gastric body is performed

SUMMARY:
Investigators assess the gastric contents by ultrasonography in fasted patients with previous subtotal gastrectomy.

DETAILED DESCRIPTION:
Investigators evaluate the gastric contents by ultrasonography in fasted patients with previous subtotal gastrectomy, quantitatively and qualitatively. The frequency of visualization fully will be also analyzed.

ELIGIBILITY:
Inclusion Criteria:

* The preoperative fasted patients with previous subtotal gastrectomy

Exclusion Criteria:

* Other anatomical abnormality or mass of stomach except gastrectomy

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will conduct a study targeting the patients with previous subtotal gastectomy among the patients fasted for an operation under general, spinal or MAC anesthesia, except people with other anatomical abnormality or mass of stomach except gastrectomy
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2018-11-15 (Actual); Primary Completion 2020-11-15 (Estimated); Study Completion 2020-12-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of full cross section image | Before the induction of anesthesia
  The gastric remnant body is assessed by ultrasound and the incidence of cross sectional image visualized fully is evaluated

SECONDARY OUTCOMES:
Type of gastric content assessed by gastric ultrasound | Before the induction of anesthesia
  The type of gastric content is assessed by gastric ultrasound; solid, fluid, empty
Cross section area of stomach body assessed by gastric ultrasound | Before the induction of anesthesia
  Cross section area is assessed by gastric ultrasound in the supine and right lateral positions
Incidence of full stomach | Before the induction of anesthesia
  It is determined if the contents is solid or the amount of fluid is large.

CONTACTS AND LOCATIONS:
Overall Officials: Tea Kyong Kim, M.D.,Ph. D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea